CLINICAL TRIAL: NCT06348355
Title: A Phase I, Open-label, Positron-Emission Tomography Study to Determine Brain Exposure of [11C]Savolitinib in Healthy Volunteers
Brief Title: A Positron-emission Tomography Study to Determine Brain Exposure of [11C]Savolitinib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D5084C00016; 2023-508334-34-00 (Other: EMA-CTIS)
Record Dates: First submitted 2024-03-12; First posted 2024-04-04 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Healthy volunteers will undergo two PET examinations and will receive 2 single IV doses of [11C]savolitinib (total ≤ 20 µg) and radioactivity of 400 ± 10% mBq/70 kg/per PET-CT examination, with total radiation exposure during the study of 3.86 mSv. Healthy volunteers will receive a single 300 mg dose of oral savolitinib approximately 2 hours after the end of the first PET examination and approximately 2 hours before the second IV dose of [11C]savolitinib. The second PET examination can be performed on a separate day, within 14 days after the first PET examination. Oral savolitinib will be given on the same day as the second PET examination.
  Interventions: Drug: [11C]savolitinib; Drug: Savolitinib

INTERVENTIONS:
Drug: [11C]savolitinib — Radiopharmaceutical; IMP; Sterile solution for IV injection, not more than 10 μg, single administration
Drug: Savolitinib — IMP; 300 mg tablet, oral single administration

SUMMARY:
The purpose of this study is to measure brain exposure of [11C]savolitinib in healthy volunteers.

This study will determine brain exposure of [11C]savolitinib in up to 8 healthy volunteers under physiological conditions, ie, when the BBB is intact. The study design allows up to 3 site visits. Two PET examinations will be performed for each healthy volunteer. The first PET examination will use IV administration of [11C]savolitinib. The second PET examination using [11C]savolitinib will occur after a single oral dose of 300 mg of savolitinib. PET image analysis will include kinetic compartment modelling using arterial input function, and will generate a set of brain exposure parameters (eg, maximum %ID, maximum [11C]savolitinib concentration in brain, partition coefficients between brain and plasma).

DETAILED DESCRIPTION:
This is a Phase I, open-label, non-randomised, single-centre study to determine brain distribution and exposure of [11C]savolitinib following IV bolus injections of a microdose in one cohort of healthy adult volunteers. The study is composed of the following parts:

Visit 1: Screening: Screening, including brain MRI, within 45 days prior to PET imaging

Visit 2: PET examination: Single microdose (≤ 10 μg) of [11C]savolitinib administered as an IV bolus at the start of PET imaging. Brain radioactivity measurements using PET/CT (radioactivity in brain) and radioactivity measurements in arterial blood (radioactivity in blood) will be taken over a maximum of 90 minutes. 300 mg savolitinib will be administered orally approximately 2 hours after the end of the first PET examination. The second microdose of [11C]savolitinib will be administered as IV bolus at approximately 2 hours after the oral administration of savolitinib, and a second PET examination will be conducted over 90 minutes. PET2 examination can be performed on a separate day, within 14 days after PET1, if it was not performed the same day due to technical/participant related reasons. Oral savolitinib will be given on the same day as the second PET examination.

Visit 3: Follow-up: Telephone assessment 7 days (± 3 days) after receiving the last microdose of [11C]savolitinib and PET examination

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers must be ≥ 50 to 65 years of age inclusive, at the time of signing the informed consent form and capable of giving informed consent.
2. Body weight within 50.0 - 100.0 kg and body mass index within the range 18.0 - 30.0 kg/m2 (inclusive).
3. Male or female with contraceptive use.

   a. Male volunteers: (i) does not wish to father any children in the 6 months after the study follow-up visit and must use condoms and spermicide with sexual partners who are pregnant or who could become pregnant from the time of dosing until 6 months after savolitinib administration.

   b. Female volunteers: Only females not of childbearing potential will be considered for enrollment in the study.

Exclusion Criteria:

1. Having known or suspected systemic infection (eg, hepatitis B virus, hepatitis C virus, human immunodeficiency virus, tuberculosis), including previous or on-going infectious or autoimmune disease.
2. Current evidence of SARS-CoV-2 infection with some exceptions applied on a case by case basis.
3. Positive urine screen for drugs of abuse at screening visit, or known history of drug or alcohol abuse within the past year.
4. Any factors that may increase the risk of QTcF prolongation such as congenital of familiar long QT syndrome, chronic hypokalemia not correctable with supplements etc.
5. Any clinically significant abnormalities on 12-lead ECG, as judged by the investigator.
6. Central nervous system infarction, infection or focal lesions of clinical significance on MRI scans.
7. Brain MRI abnormalities that would interfere with image analysis, as determined by the PI
8. Presence of significant abnormalities in the medical history or physical examination or laboratory tests at screening that may interfere with the study or present a safety risk.
9. Current significant major or unstable respiratory, heart, cerebrovascular, haematological, hepatic, renal, gastrointestinal diseases, or other major disease.
10. Any concomitant medications known to be associated with Torsades de Pointes, potent inducers of cytochrome P450 3A4 (CYP3A4), strong inhibitor of CYP1A2, inhibitors or inducers of P-gp.
11. Participation in a research PET or PET/CT study in the previous 12 months, and as per the judgement of the PI participation in this study will not expose the volunteer to radiation in excess of internationally accepted limit.
12. History of autoimmune disease, severe/ongoing allergy or atopy, or history of hypersensitivity to drugs with a similar chemical structure or class to [11C]savolitinib/savolitinib or the excipients of [11C]savolitinib/savolitinib.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Percentage of injected radioactivity entering the brain (%ID) as %IDmax_brain | 0-90 minutes post IV dose of [11C]savolitinib
  Determine brain exposure of [11C]savolitinib following single, IV administration of a microdose in healthy adult volunteers

SECONDARY OUTCOMES:
The following endpoint: Cmax_brain SUV | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single, IV administration of a microdose
The following endpoint: Tmax brain | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single, IV administration of a microdose
The following endpoint: AUCbrain 0-90 | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single, IV administration of a microdose
The following endpoint: AUCplasma 0-90 | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single, IV administration of a microdose
The following endpoint: Kp | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single, IV administration of a microdose
The following endpoint: Kp,uu | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single, IV administration of a microdose
The following endpoint: VT | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single, IV administration of a microdose
The following endpoint: Cmax_brain SUV | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single oral dose of 300 mg of savolitinib
The following endpoint: Tmax brain | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single oral dose of 300 mg of savolitinib
The following endpoints: AUCbrain 0-90 | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single oral dose of 300 mg of savolitinib
The following endpoints: AUCplasma 0-90 | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single oral dose of 300 mg of savolitinib
The following endpoints: Kp | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single oral dose of 300 mg of savolitinib
The following endpoints: Kp,uu | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single oral dose of 300 mg of savolitinib
The following endpoints: VT | 0-90 minutes post IV dose of [11C]savolitinib
  Estimate brain exposure of [11C]savolitinib in healthy adult volunteers after single oral dose of 300 mg of savolitinib

OTHER OUTCOMES:
Number of participants with safety findings, AEs | Through study completion, up to 69 days (including screening period)
  Provide additional safety and tolerability information for [11C]savolitinib IV and savolitinib oral administration (single dose)

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Svensson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Research Site, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5084C00016&attachmentIdentifier=e110ee4e-4001-4ca2-804b-d4901d6164fc&fileName=d5084c00016-study-synopsis_Redacted_final_(1).pdf&versionIdentifier=